CLINICAL TRIAL: NCT06353854
Title: National French Cohort Evaluating Predictive Factors of Resistance to Immunotherapy in Patients With MSI Metastatic Colorectal Cancer
Brief Title: Prospective National Cohort Evaluating Predictive Biomarkers of Resistance to Immunotherapy in Patients With MSI/dMMR Metastatic Colorectal Cancer (CORESIM)
Acronym: CORESIM
Status: Recruiting | Type: Observational
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Other Study IDs: FFCD 2112-CORESIM
Record Dates: First submitted 2024-03-28; First posted 2024-04-09 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Colorectal Cancer Metastatic; Microsatellite Instability-High Colorectal Cancer
Keywords: immunotherapy resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Tumor samples archived for retrospective cohort Tumour samples archived and blood samples at 3 time points for prospective cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Retrospective group: Registration of patients treated with pembrolizumab since February 2021. Collection of tumour sample archives will be associated
- Prospective group: Recruitment of metastatic colorectal cancer patients with microsatellite instability prior to the first administration of pembrolizumab immunotherapy. Blood and tumour sampling will be combined.

SUMMARY:
The Keynote 117 phase III trial demonstrated the superiority of pembrolizumab (anti-PD1 monoclonal antibody) versus chemotherapy +/- targeted therapy in first-line treatment of dMMR/MSI metastatic colorectal cancer (mCRC). However, primary resistance to pembrolizumab was observed in approximately 20-30% of patients treated in the Keynote 177 study. Therefore, the identification of biomarkers predictive of resistance to immunotherapy for dMMR/MSI mCRC is necessary to better select patients who benefit the most from immunotherapy, and those for whom other therapeutic approaches should be favored.

DETAILED DESCRIPTION:
The primary endpoint is the identification of predictive factors of resistance to pembrolizumab in first-line treatment of MSI and/or dMMR metastatic colorectal cancer

CORESIM is a retrospective and prospective multicenter national French cohort. National recruitment will be carried out in all French centers, including the FFCD, AGEO, GERCOR, and UNICANCER, representing more than 150 centers and most French sites, public and private hospitals.

In France, pembrolizumab for first-line treatment of patients with MSI mCRC was accessible via its compassionate use in February 2021, then its reimbursement was effective in June 2023 Patients treated with pembrolizumab will be included prospectively on the start date of the study, i.e. on February 2024; patients treated since February 2021 via compassionate use of pembrolizumab will be included retrospectively A total of 600 patients are expected. The theoretical duration of inclusion is set at 2 years. All patients will be followed up for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Histologically confirmed colorectal adenocarcinoma with unresectable metastasis(s) receiving immunotherapy as first-line treatment with pembrolizumab
* Tumor with microsatellite instability determined by immunohistochemistry (loss of expression of MLH1, MSH2, MSH6 and/or PMS2) and/or by molecular biology (MSI-H on microsatellite analysis from tumor DNA according to practice routine of the center)

Exclusion Criteria:

* Patients with another concomitant cancer at the time of diagnosis requiring systemic treatment or impacting prognosis according to the medical team.
* Previous treatment with anti-PD1 or anti-PDL1.
* Previous treatment with chemotherapy +/- targeted therapy for MSI/dMMR metastatic colorectal cancer.
* Contraindication due to psychological or social reasons that may hinder follow-up (cognitive deficit, psychological disorders incompatible with obtaining non-opposition or consent; inability to be followed in the same center throughout the follow-up period for geographical reasons).
* Pregnant women
* persons under court protection or under protective supervision (guardianship or curatorship)
* Opposition to participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective inclusion of patients receiving first-line immunotherapy with pembrolizumab (as defined in the MA) for unresectable mCRC.
  Patients who have received pembrolizumab in the same indication on a compassionate basis since February 2021 may also be retrospectively included in the cohort.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2029-02-12 (Estimated); Study Completion 2030-02-12 (Estimated)

PRIMARY OUTCOMES:
Identification of predictive factors of resistance to pembrolizumab in first-line treatment of MSI and/or dMMR metastatic colorectal cancer | 2 years
  Primary resistance will be defined as immediate progression of the disease (at the time of the first assessment, excluding pseudoprogression) Secondary resistance will be defined as progression occurring after control of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Aziz ZAANAN, MD, PhD, Principal Investigator — Hôpital Européen Georges Pompidou APHP
Locations (20):
- France (20):
  - Ch - Centre Hospitalier de La Côte Basque, Bayonne
  - Ch - Ch Beauvais, Beauvais
  - CH Jean Minjoz, Besançon
  - Polyclinique Saint Privat, Boujan-sur-Libron
  - Ch - Duchenne, Boulogne-sur-Mer
  - Ch - Centre Hospitalier Metropole Savoie, Chambéry
  - Ch - Centre Hospitalier de Cholet, Cholet
  - CH - Compiegne, Compiègne
  - Ch - Chd Vendée, La Roche-sur-Yon
  - CH - Louis Pasteur, Le Coudray
  - Centre Hospitalier Regional et Universitaire de Lille, Lille
  - CH Saint Joseph - Saint Luc, Lyon
  - Caluire et Cuire - Infirmerie Protestante de Lyon, Lyon
  - Ch - Hôpital Saint Joseph, Marseille
  - CH Saint Joseph, Marseille
  - Centre Hospitalier, Mulhouse
  - CHR D'Orleans - Hopital de la Source, Orléans
  - Prive - Institut Montsouris, Paris
  - Ch - Centre Hospitalier de Soisson, Soissons
  - CH - Gustave Dron, Tourcoing